CLINICAL TRIAL: NCT00619125
Title: A Proposal to Evaluate Time-specific Relationships Between Variables of Pain, Stress, and Bloating in the Onset of IBS Diarrhea and Constipation Symptoms Using Ecological Momentary Assessment (EMA)
Brief Title: Proposal Evaluating Time-specific Relationships Between Variables of Pain, Stress, and Bloating in IBS Diarrhea and Constipation Symptoms Using a Palm Pilot
Status: Completed | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Takeda Pharmaceuticals North America, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 07-1782
Record Dates: First submitted 2008-01-24; First posted 2008-02-20 (Estimated); Last update posted 2017-06-20 (Actual); Status verified 2011-10

CONDITIONS: IBS, Diarrhea Predominant; IBS, Constipation Predominant; IBS, Mixed Symptoms
MeSH Terms: conditions — Ichthyosis Bullosa of Siemens

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- A: 20 patients with IBS C
  Interventions: Other: palm pilot recording responses to questionnaires
- D: 20 Subjects without IBS
- B: 20 patients with IBS D
  Interventions: Other: palm pilot recording responses to questionnaires
- C: 20 patients with IBS M
  Interventions: Other: palm pilot recording responses to questionnaires

INTERVENTIONS:
Other: palm pilot recording responses to questionnaires — Short interval assessment (provided by data from palm pilot) may provide a more accurate picture of patient symptom experience.
  Groups: A; B; C

SUMMARY:
Purpose: The associations between pain, stress, bloating, and their short interval temporal relationships to defecation in IBS D, C & M are of great interest to the field of functional GI disorders, but have not been adequately studied. Broad recall based assessments (i.e.,over past week or month) of pain and bloating have been key features of the diagnosis of IBS, however such long term retrospective recall of symptom experience has been shown to be unreliable and influenced by outside factors (heuristics, recall bias, etc.). Short interval assessment may provide a more accurate picture of patient symptom experience Participants: Patients with IBS in general and IBS subtypes (IBS-C, D, M) Procedures (methods): Study participants could be asked to record data at randomly assigned points throughout the day, as well as during the course of a diarrheal or constipated stool (i.e., prior to and right after a bowel movement).

ELIGIBILITY:
Inclusion Criteria:

1. The subject signs and dates a written informed consent form (ICF) prior to any study-related activities, including discontinuation of any prohibited medications.
2. The subject has been diagnosed with either IBS-C, IBS-D, IBS-M, or has no history of gastrointestinal symptoms (control group).
3. The subject has at least 3 pain episodes a week and does not have constant, unremitting abdominal pain.
4. The subject is at least 18 years of age and less than 75 years of age at the time of the screening visit.
5. The subject is fluent in English.
6. The subject is an ambulatory outpatient. Ambulatory is defined as not depending exclusively on a wheelchair for mobility. Nursing home subjects may be enrolled provided they are ambulatory. Subjects with spinal cord injuries resulting in paraplegia may not be enrolled.

Exclusion Criteria:

1. The subject exhibits evidence of a biochemical or structural abnormality of the digestive tract. These conditions include (but are not limited to) the following:

   * Inflammatory bowel disease (Crohn's disease or ulcerative colitis),
   * GI surgery (with the exceptions of appendectomy; cholecystectomy; benign polypectomy; fundoplication without gas bloat syndrome, 6 months post-surgery; herniorrhaphy without bowel resection, 1 month post-surgery; hemorrhoidectomy, at least 2 months post-surgery; and hiatal hernia repair),
   * GI malignancy, GI obstruction
2. In the opinion of the investigator the subject has a concurrent illness or disability (excluding IBS) that may affect the interpretation of clinical efficacy and/or safety data or otherwise contraindicates participation in this clinical study (e.g., an unstable cardiovascular, renal, hepatic, pulmonary, endocrine, metabolic, GI, hematological, or neurological condition).
3. The subject has been diagnosed with a major psychiatric disorder within the past 2 years that required hospitalization and/or involved an attempted suicide (e.g., major depression or psychoses). Subjects diagnosed with a major psychiatric disorder that did not require hospitalization or involve an attempted suicide must have remained on a stable dose of medication for at least 6 months prior to the screening visit.
4. The subject has a history of alcohol or substance abuse within the past 2 years.
5. The subject has any evidence or treatment of malignancy (other than localized basal cell, squamous cell skin cancer or cancer in situ that has been resected) within the previous 5 years.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 80 male and female subjects will be recruited: 20 with IBS D; 20 with IBS C; 20 with IBS M; 20 control (no bowel symptoms).
  We will target patients who have maintained a diagnosis of IBS with Diarrhea (IBS-D), IBS with Constipation (IBS-C, IBS with Mixed Stool pattern (IBS-M), using Rome III Criteria as well as control subjects without bowel symptoms. Subject participation will be limited to patients who maintain mild or moderate symptom severity score on the functional bowel disorders severity index (FBDSI.) providing they have at least 3 symptom episodes of pain or discomfort in a given week, to assure adequate data collection.
Sampling Method: Probability Sample
Enrollment: 85 (Actual)
Dates: Start 2008-04; Primary Completion 2009-03 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
To determine relation of pain and bloating relative to average pain and bloating scores | 2 weeks

SECONDARY OUTCOMES:
determine the association of acute stress with increased pain and bloating scores or with defecation in IBS | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Douglas Drossman, MD, Principal Investigator — UNC-Chapel Hill